CLINICAL TRIAL: NCT04390256
Title: Remineralization of Early Carious Lesion Using Natural Agents Versus Bioadhesive Polymers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed, Ass. lecturer, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC17-030
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — carboxypolymethylene

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Egg shell powder nanoparticles (Active Comparator)
  Interventions: Other: Clove water extract; Other: Carbopol; Other: Carboxymethyle cellulose
- Clove water extract (Experimental)
  Interventions: Other: Clove water extract; Other: Carbopol; Other: Carboxymethyle cellulose
- Carbopol (Experimental)
  Interventions: Other: Clove water extract; Other: Carbopol; Other: Carboxymethyle cellulose
- Carboxymethyle cellulose (Experimental)
  Interventions: Other: Clove water extract; Other: Carbopol; Other: Carboxymethyle cellulose

INTERVENTIONS:
Other: Clove water extract — natural product
Other: Carbopol — Bioadhesive polymer
Other: Carboxymethyle cellulose — Bioadhesive polymer

SUMMARY:
This study will be conducted to evaluate:

1. The remineralization potential of natural agents (egg shell powder and clove extract) versus bioadhesive polymers (carbopol and carboxymethyl cellulose) with or without PH cycling using microhardness test.
2. The clinical efficacy of all agents in patients with early carious lesions.

ELIGIBILITY:
Inclusion Criteria:

* 1. Criteria related to patient:

  * Age's eligible for trial was 18- 30 years.
  * Patient able to read and sign the informed consent form.
  * Cooperative patient who are willing to participate and able to continue the schedule time of wok keep good oral hygiene throughout the study.
  * Healthy volunteers.
  * Patient with moderate and high caries index. 2. Criteria related to tooth:
  * Patient with at least 2 white lesions (WSL) detected clinically on the buccal surface of permanent anterior teeth, one on each side. WSL selected either due to caries or orthodontic treatment (just following deboning).
  * Teeth with score1, 2, 3 according to ICDAS II.
  * Absence of preoperative pain, no mobility & tenderness on percussion.
  * Radiographically, the pre-operative inclusion criteria were absence of internal or external resorption, no periapical radiolucencies and no widening of periodontal ligament space..

Exclusion Criteria:

* 1. Criteria related to patient:

  * Patient with Rampant uncontrolled caries.
  * Patient with compromised medical history.
  * Pregnant or breast feeding females.
  * Heavy smoker.
  * Patient who currently received extensive fluoride regiments for treatment of WSL.
  * Patients who planned to move within 3 months of enrollment.
  * Patient with evidence of xerostomia. 2. Criteria related to tooth:
  * Teeth with score 4, 5 according to ICDAS II.
  * Teeth with periapical pathology, internal or external resorption or exhibiting any symptoms of pulp pathology.
  * Teeth with questionable vitality or have root canal therapy.
  * Teeth have been pulp capped.
  * Teeth with periodontal pocket and bleeding on probing.
  * Cracked teeth.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Remineralization of enamel | 3 months
  Remineralization of enamel using Vista scan

CONTACTS AND LOCATIONS:
Locations (1):
- Al Azhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided